CLINICAL TRIAL: NCT06660056
Title: A Phase I Study Evaluating the Safety, Tolerability, Biodistribution and Shedding of Oncolytic Vaccinia Virus GC001, Pharmacodynamics, Immunogenicity, and Antitumor Activity of the Virus in Patient With Recurrent or Progressive Gliomas
Brief Title: A Phase I Clinical Study of Intratumoral Injection GC001 in Patient With Recurrent or Progressive Gliomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GONGCHU Biotechnology Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GONGCHU Bio
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-10

CONDITIONS: High-grade Gliomas
Keywords: Oncolytic virus; GC001; WR; high-grade gliomas

STUDY DESIGN:
Intervention Model Description: 3+3
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): The study consists of a total of seven dose groups, with the lowest dose group being 1×10^6 and the highest dose reaching 1×10^9 PFU.To avoid exposing too many subjects to an ineffective dose, accelerated titration will be used for the 1 x 10^6 pfu and 3 x 10^6 pfu dose groups. The 1×10^7-1×10^9 pfu dose group will be dose-escalated using the traditional "3+3" design. In case the maximum dose of 1×10^9 PFU fails to achieve the Maximum Tolerated Dose (MTD), the sponsor and the investigator will convene to discuss whether to designate it as Maximum Feasible Dose (MFD) or consider escalating further based on current safety and preliminary efficacy data. However, any escalation beyond that of similar drugs' Phase I clinical trials, such as JX-594:NCT00629759 and JX-929:NCT00574977, where the highest administered dose was 3×10^9 PFU, shall be avoided. This precaution ensures adherence to established safety protocols.
  Interventions: Biological: A Phase I Clinical Study of Intratumoral Injection Oncolytic Vaccinia Virus GC001 in Patient With Recurrent or Progressive Gliomas of the Brain
- Part 2:metrological amplification stage (Experimental): Based on the MTD determined during the dose-escalation phase (or the investigator's or sponsor's assessment to select a more appropriate dose), patients with recurrent or progressive gliomas who standard therapy failure or intolerance will be included, and will be enrolled 10 to 30 subjects.
  Interventions: Biological: A Phase I Clinical Study of Intratumoral Injection Oncolytic Vaccinia Virus GC001 in Patient With Recurrent or Progressive Gliomas of the Brain

INTERVENTIONS:
Biological: A Phase I Clinical Study of Intratumoral Injection Oncolytic Vaccinia Virus GC001 in Patient With Recurrent or Progressive Gliomas of the Brain — Use of Ommaya capsules

SUMMARY:
A Phase I Study Evaluating the Safety, Tolerability, Biodistribution and Shedding of the Virus, Pharmacodynamics, Immunogenicity, and Antitumor Activity of GC001 Oncolytic Vaccinia Virus Injection in Patient With Recurrent or Progressive Gliomas .

DETAILED DESCRIPTION:
The ongoing trial is structured as an open, single-arm Phase I clinical study consisting of dose-escalation and dose-expansion.

The main objective of dose-escalation is:

To evaluate the safety and tolerability i.e. dose limiting toxicity (DLT), maximum tolerated dose (MTD) or maximum administered dose (MFD) of GC001 injection in patients with with recurrent or progressive gliomas,and will be determining the recommended phase II dose(PR2D).

The initial phase of the study, Part I, utilizes a 3+3 design to meticulously evaluate the escalation of the dose of GC001. The total enrollment of participants will be determined by the observed toxicity levels and the extent of dose cohorts explored, with a maximum enrollment of 42 cases. A critical 28-day period post-administration has been established for the observation of dose-limiting toxicities (DLTs) to ensure participant safety. It is essential to maintain this standardized 28-day observation window for all enrolled groups to uphold the highest safety standards.

The secondary aims of this dose-escalation are to assess the biodistribution and shedding of the virus, the pharmacodynamic characteristics, immunogenicity, and the initial antitumor efficacy of the GC001 injection in patients suffering from advanced with recurrent or progressive gliomas.

Following the completion of the DLT assessment for all participants within each dose cohort, the SMC may decide whether to proceed with dose escalation, explore intermediate/higher doses, or terminate the dose escalation study based on the data obtained on safety, tolerability, biodistribution, and shedding of the virus (if any), pharmacodynamics (if any), immunogenicity (if any), and antitumor activity (if any). The SMC may also decide to adjust doses, administration schedules, and the time of biospecimen collection.

To further evaluate the safety and preliminary antitumor activity of GC001 Oncolytic Vaccinia Virus Injection in the treatment of patients with With recurrent or progressive gliomas during the dose-expansion phase.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for participation in this study, individuals must meet the following criteria:

1. Subjects must be able to comprehend and voluntarily sign written informed consent, which includes requirements related to study sample collection.
2. Able to communicate with researchers; Understand and comply with the requirements of the study; Voluntary and able to complete study procedures and follow-up examinations.
3. Be male or female patients aged 18 (including those with borderline age values).
4. Patients with recurrent or progressive high-grade gliomas (WHO grade III-IV) that have been histopathologically or molecularly diagnosed and for which there is either no current standard of care or the standard treatment has proven ineffective (progression of the disease after treatment or intolerance of treatment).
5. At least 1 intracranial measurable lesion according to RANO criteria (well-defined enhancing lesion detected on MRI, diameter >10 mm).
6. Patient's willingness to undergo surgical maneuvers related to placement of the Ommaya capsule.
7. Karnofsky functional status ≥ 60.
8. Be expected to survive for at least 3 months.
9. No serious hematologic (no adjuncts such as EPO, G-CSF, or GM-CSF within 14 days prior to the first dose and no blood transfusions for at least 7 days), hepatic, or renal function abnormalities consistent with the following laboratory test results:

systems Laboratory test values routine blood test Absolute neutrophil count（ANC） ≥1.5×109/L blood platelet（PLT） ≥100×109/L hemoglobin（HGB） ≥90g/L gallbladder serum creatinine（Cr） ≤1.5×Upper limit of normal range（ULN） creatinine clearance（Ccr）（To be calculated only if creatinine > 1.5 x ULN） ≥50mL/min（Based on the Cockcroft-Gault formula） liver total bilirubin（TBIL） ≤1.5×ULN glutamic pyruvic transaminase（ALT） aspartate transaminase（AST） ≤2.5×ULN Alkaline phosphatase（ALP） ≤2.5×ULN coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5×ULN Partially activated thromboplastin time（APTT） ≤1.5×ULN 10.Male or female subjects of childbearing potential use effective contraception during treatment and for 6 months after dosing.

Exclusion Criteria:

1. Inability to perform an MRI for any reason.
2. focal point under the curtain.
3. Prior history of encephalitis, multiple sclerosis, or other central nervous system infection (unless resolved).
4. Patients with a previous diagnosis of any other malignancy within 5 years prior to the first dose, except for malignancies with a low risk of metastasis and risk of death (5-year survival > 90%), such as adequately treated basal cell or squamous cell skin cancer, cervical carcinoma in situ, and other carcinomas in situ.
5. Females of childbearing age who have a positive pregnancy test or are lactating.
6. Individuals with allergies (defined as ≥2 drug allergies) or hypersensitivity to similar products or excipients.
7. Those who have received smallpox vaccination and experienced severe systemic reactions or side effects.
8. Patients who have previously received lysosomal virus, stem cell, or gene therapy products.
9. Individuals using other investigational drugs or participating in clinical trials of other drugs within 28 days prior to the first dose (except for those who did not receive the test drug).
10. Those who have undergone antitumor therapy, including radiation therapy (except palliative radiotherapy), chemotherapy, biotherapy, endocrine therapy, and immunotherapy within 28 days prior to the first administration of the drug.
11. Individuals who have undergone surgery or interventional therapy (excluding tumor biopsy, puncture, Ommaya capsule etc.).
12. Individuals who have been treated with systemic corticosteroids (at a dose equivalent to >10 mg dexamethasone /day) or other immunosuppressive medications within 28 days prior to the first dose, or who are currently taking antiviral medications (Mainly sensitive to poxviruses), enrollment is permitted under the following cases:

    1. short-term (≤7 days) use of corticosteroids for prophylaxis or treatment of non-autoimmune allergic diseases is permitted;
    2. the use of topical topical or inhaled glucocorticoids is permitted;.
13. A history of severe cardiovascular disease, including but not limited to:

    1. A history of severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias, degree II-III AV block requiring clinical intervention;
    2. Acute coronary syndrome, congestive heart failure, aortic coarctation, stroke, or other grade or greater cardiovascular event within 6 months prior to the first dose;
    3. New York Heart Association (NYHA) > Class II heart failure or left ventricular ejection fraction (LVEF) <50%; heart rate-corrected baseline QTcF intervals >450msec (men) and >470msec (women) using the Fridericia formula; any factor that increases the risk of QTc prolongation or the risk of cardiac arrhythmias, such as heart failure, hypokalemia , congenital long QT syndrome, family history of long QT syndrome, or use of any concomitant medication known to prolong the QT interval；
    4. Clinically uncontrolled hypertension (blood pressure uncontrolled at < 160 mmHg systolic and < 100 mmHg diastolic after standard antihypertensive treatment).
14. Recent Grade 3 or greater bleeding event within 6 months prior to the first use of study drug, or who have current > Grade 2 bleeding, or hemangioma/vascular malformation, or tumor stroke, tumor invasion of a blood vessel, or active peptic ulcer, or esophageal varices judged by the investigator to be at significant risk for bleeding.
15. Those with a history of severe hemoptysis.
16. Patients with uncontrolled or severe diseases, including but not limited to persistent or active infections requiring antibiotic therapy.
17. .Subjects with active or prior history of autoimmune diseases with potential for recurrence (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulonephritis, etc.) or at high risk (e.g., patients who have undergone organ transplantation requiring immunosuppressive therapy) are not eligible for enrollment. However, enrollment is permitted for subjects with:

    1. type 1 diabetes mellitus that is stabilized on a fixed dose of insulin;
    2. autoimmune hypothyroidism or Hashimoto's thyroiditis that requires only hormone replacement therapy；
    3. Individuals with a history of exfoliative skin conditions requiring systemic therapy (e.g., eczema or atopic dermatitis) are also excluded.
18. Persons who are positive for human immunodeficiency virus (HIV) antibodies.
19. Persons who have active hepatitis B (HBV)/hepatitis C (HCV) infection are not eligible for enrollment. However, subjects with a previous history of hepatitis C but negative HCV RNA at screening may be enrolled, and those who are HBsAg positive but have HBV DNA <500 IU/ml or below the lower limit of detection at the study center may also be enrolled. Subjects with primary liver cancer and HBV DNA <1000 IU/ml may be enrolled as well.
20. Patients with documented psychiatric illnesses or disorders that may impact adherence to the trial protocol.
21. Patients with malignant tumors that may require antitumor therapy other than the investigational drug GC001.
22. Patients who, as determined by the investigator, are unsuitable for participation in the study.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-02-08 (Estimated); Study Completion 2026-08-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of GC001 | DLT Observation Period，Up to 28 days from GC001 injection
  Number of participants in dose escalating cohorts with dose limiting toxicities (DLTs)，treatment-emergent adverse events (TEAEs), and/or changes in clinical laboratory abnormalities.
Maximal tolerable dose | DLT Observation Period,Up to 28 days from GC001 injection
  During the DLT observation period, the number of cases with DLT is less than or equal to the maximum dose of 1/6 of the total number of cases, and six evaluable participants are required to determine MTD.

SECONDARY OUTCOMES:
Anti-tumor activity of GC001: response assessment of neuro-oncology(RANO). | Up to 2 years
  To evaluate the response assessment of neuro-oncology(RANO) as a measurement of tumor response and disease progression.
Anti-tumor activity of GC001: immunotherapy response assessment for neuro-oncology (iRANO). | Up to 2 years from GC001 injection
  To evaluate the immunotherapy response assessment for neuro-oncology (iRANO) as a measurement of tumor response and disease progression.

OTHER OUTCOMES:
Evaluate the viral biological distribution and shedding of GC001 | Up to 2 years from GC001 injection
  Viral biodistribution and shedding analysis for GC001 injection are performed based on the viral Biodistribution and shedding Analysis Set (BVSS). Biological collection samples include blood, urine, throat swabs, omaya cyst aqueous ,injection site and injection site dressing samples (for tumor injection at the percutaneous puncture site only),and determination of viral DNA copy number in the above samples.
Pharmacodynamic analysis of cytokine levels in the peripheral blood and omaya cyst aqueous. | Up to 2 years from GC001 injection
  To assess the levels of cytokines including IFN-γ, TNF-α, IL-5、 IL-6 and IL-10 in the peripheral blood andomaya cyst aqueous.
Pharmacodynamic analysis of PD-1 and lymphocyte in the peripheral blood and omaya cyst aqueous | Up to 2 years from GC001 injection
  To assess the ratio of PD-1 and lymphocyte in the peripheral blood and omaya cyst aqueous.
immunogenicity | Up to 2 years from GC001 injection
  Immunogenicity analysis will measure the concertation of antidody (anti-VV antibody (ADA) and neutralizing antibody (Nab) )in the peripheral blood.
Pharmacodynamic analysis of immune cells in the peripheral blood and omaya cyst aqueous | Up to 2 years from GC001 injection
  The lymphocyte ratio of CD3 + / CD4 + , CD3 + / CD8 + and the ratio of CD4 + / CD8 + are measured in the peripheral blood and omaya cyst aqueous.

CONTACTS AND LOCATIONS:
Overall Officials: li gongchu, Professor, Principal Investigator — GONGCHU Biotechnology Co., Ltd
Locations (1):
- Beijing Tiantan Hospital,Capital Medical University, Beijing, Beijing Municipality, China